CLINICAL TRIAL: NCT04885075
Title: A Randomized Controlled Trial Comparing the Efficacy of Intranasal Midazolam and Conventional Treatment With Intravenous Diazepam for Control of Seizures in Children
Brief Title: Comparing the Efficacy of Intranasal Midazolam Versus Intravenous Diazepam for Control of Seizures in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr Nighat Haider, assistant professor of paediatrics, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.F.1-1/2015/ERB/SZABMU/602
Record Dates: First submitted 2021-03-28; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Diazepam; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Diazepam (Other): Intravenous diazepam (0.2mg/kg/dose) single dose stat
  Interventions: Drug: IV diazepam
- Intranasal Midazolam (Other): Intranasal midazolam (0.2mg/kg/dose) single dose stat
  Interventions: Drug: I/N Midazolam

INTERVENTIONS:
Drug: IV diazepam — inj.diazepam 0.2mg/kg/dose stat
  Other Names: valium
  Arms: Intravenous Diazepam
Drug: I/N Midazolam — intranasal midazolam 0.2mg/kg/dose stat
  Other Names: dormicum
  Arms: Intranasal Midazolam

SUMMARY:
After approval , study will be conducted at the Children Hospital PIMS, Islamabad. Children 1-12 years presenting/admitted with seizures will be enrolled in the study after taking informed consent from the parents. Children's name, age, sex will be recorded by the on duty doctor. Patients will be randomly allocated to two equal groups. Group A (GA) will receive single dose of intravenous diazepam (0.2mg/kg/dose)after passing cannula, while Group B (GB) will receive single dose of intranasal midazolam (0.2mg/kg/dose).Response to treatment will be assessed by recording the time required for termination of seizures in both gruops.the time required for gaining intravenous accessin Group A will be recorded as well. Data will be collected through a structured performa.

DETAILED DESCRIPTION:
Benzodiazepines are the first line of drugs for cessation of acute seizures.benzodizepines can be given intravenous,orally,per rectal and intranasal.Conventional treatment of acute seizures is intravenous diazepam in most hospital settings which requires an IV access,which is not possible for parents to give at home.The main problem in an actively seizuring child is to reach the hospital and maintaining an intravenous line.Midazolam is a water soluble benzodiazepine which is widely used as an anxiolytic and anticonvulsant ,can be given through intravenously,intramuscularly, oral,buccal and nasal mucosa as well.it becomes lipid soluble at physiologic PH levels and reaches the CNS with a rapid onset and shorter duration of action.It is administered into nostril in a way that it comes into direct contact with nasal mucosa.It is given in a dose of 0.2mg\kg and within a few minutes its level in serum are comparable to the injectables levels.It is a safe,cheap,easy to use and effective alternative to diazepam for use at home as well as in hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-10 years both male and female visiting/admitted in Children Hospital PIMS with acute episode of seizure (febrile or afebrile)

Exclusion Criteria:

* Children requiring emergency resuscitation
* Children with uncontrolled epilepsy

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-05-30 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Time taken for seizures to be controlled | From administration of drug to the cessation of seizures up to 10 minutes
  Intranasal midazolam will take less time for cessation of seizure than intravenous diazepam

CONTACTS AND LOCATIONS:
Overall Officials: nighat haider, mbbs,fcps, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University

IPD SHARING:
Plan to Share IPD: No